CLINICAL TRIAL: NCT03430180
Title: Double-blind, Placebo-controlled Randomised Study on the Efficacy of Naloxone Nasal Spray for the Treatment of Gambling Disorder
Brief Title: Effects of Intranasal Naloxone on Gambling Urges and Craving in Gambling Disorder
Acronym: NalGamb
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Hannu Alho, Research professor, Finnish Institute for Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NalGamb; 2017-001946-93 (EudraCT Number)
Record Dates: First submitted 2018-01-30; First posted 2018-02-12 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Pathological Gambling; Gambling Disorder; Opioid Antagonist; Naloxone
MeSH Terms: conditions — Gambling | interventions — Naloxone

STUDY DESIGN:
Intervention Model Description: Treatment Group A: Naloxone hydrochloride 40mg/ml nasal spray Naloxone hydrochloride will be dosed at 4mg / dose (one spray of 0.1ml of the 40mg/ml formulation into one nostril) up to four times daily as needed in response to gambling urges with at least 2 hours between each dose (within 24 hours from 6am each day) for 12 weeks.
  One spray of naloxone hydrochloride 40mg/ml nasal spray contains 4 mg naloxone hydrochloride in a formulation of benzalkonium chloride, sodium edetate, sodium chloride, hydrochloric acid and purified water.
  Treatment Group B: Placebo nasal spray One spray of 0.1ml of the placebo formulation in one nostril up to four times daily as needed in response to gambling urges with at least 2 hours between each dose (within 24 hours from 6am each day) for 12 weeks.
  One spray of placebo nasal spray contains benzalkonium chloride, sodium edetate, sodium chloride, hydrochloric acid and purified water
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- placebo nasal spray (Placebo Comparator): Drug: placebo nasal spray One spray of 0.1ml of the placebo formulation in one nostril up to four times daily as needed in response to gambling urges with at least 2 hours between each dose (within 24 hours from 6am each day) for 12 weeks.
  Interventions: Drug: Placebo
- Naloxone hydrochloride 40mg/ml nasal spray (Active Comparator): Naloxone hydrochloride will be dosed at 4mg / dose (one spray of 0.1ml of the 40mg/ml formulation into one nostril) up to four times daily as needed in response to gambling urges with at least 2 hours between each dose (within 24 hours from 6am each day) for 12 weeks.
  Interventions: Drug: Naloxone hydrochloride

INTERVENTIONS:
Drug: Naloxone hydrochloride — Naloxone hydrochloride will be dosed at 4mg / dose (one spray of 0.1ml of the 40mg/ml formulation into one nostril) up to four times daily as needed in response to gambling urges with at least 2 hours between each dose (within 24 hours from 6am each day) for 12 weeks.
  Other Names: Naloxone 40mg/ml nasal spray when craving to gamble
  Arms: Naloxone hydrochloride 40mg/ml nasal spray
Drug: Placebo — One spray of 0.1ml of the placebo formulation in one nostril up to four times daily as needed in response to gambling urges with at least 2 hours between each dose (within 24 hours from 6am each day) for 12 weeks.
  Other Names: Placebo nasal spray with no active ingredients
  Arms: placebo nasal spray

SUMMARY:
Primary objective:

*To determine whether treatment with naloxone hydrochloride nasal spray reduces gambling urge symptoms in patients with gambling disorder

The secondary objectives of the study are:

* To determine the effects of naloxone hydrochloride nasal spray on gambling severity, frequency and time, internet use, self-efficacy, quality of life, alcohol consumption, depression
* To evaluate the safety of naloxone hydrochloride nasal spray in the treatment of gambling disorder

DETAILED DESCRIPTION:
This is a 12 week, randomised, double-blind, placebo-controlled, parallel group study to determine the efficacy of naloxone hydrochloride nasal spray in gambling disorder. Anticipated number of participants are 126.

Treatment Group A: Naloxone hydrochloride 40mg/ml nasal spray Naloxone hydrochloride will be dosed at 4mg / dose (one spray of 0.1ml of the 40mg/ml formulation into one nostril) up to four times daily as needed in response to gambling urges with at least 2 hours between each dose (within 24 hours from 6am each day) for 12 weeks.

Treatment Group B: Placebo nasal spray One spray of 0.1ml of the placebo formulation in one nostril up to four times daily as needed in response to gambling urges with at least 2 hours between each dose (within 24 hours from 6am each day) for 12 weeks.

Safety parameters:

Study Subjects will be asked to report any changes in health via the daily questionnaire. This will be reviewed weekly and at each study Visit (including phone calls) and any adverse events will be documented in the eCRF. Changes in vital signs and outcome of routine blood analyses will be evaluated.

Adverse events (AEs) will be classified using a coding thesaurus (MedDRA).

Primary endpoint: Gambling symptoms (G-SAS) from Baseline to week 12. Gambling symptoms (G-SAS) from Baseline to week 12.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

The Subject must satisfy the following criteria for entry into the study:

1. Aged 18 to 75 years, fluent in Finnish and able to read and understand the patient information sheet
2. Provide written, informed consent prior to any study specific procedure being conducted
3. Gambling problem at pre-screening (SOGS 5 or more points)
4. Moderate (6-7 criteria met) or severe (8-9 criteria met) GD (DSM-5) assessed by clinical interview with Medical Doctor (MD)
5. At least 4 weeks since completion of any other previous treatment for GD
6. At least 8 weeks since completion of any previous treatment with naltrexone or nalmefene
7. Willingness to comply with all study procedures and visit schedules

Exclusion Criteria:

* Exclusion criteria:

The Subject will be excluded from the study if any of the following applies:

1. Two weeks or longer abstinence from gambling prior to randomisation
2. Known allergic reactions to naloxone or excipients of IMP and placebo
3. Current use of drugs (opiates, amphetamine, metamphetamine, cocaine, cannabis and benzodiazepines) (as assessed by saliva drug screen, DrugWipe-6)
4. Subject is taking any prohibited medication (opioid analgesics, any medication delivered to the nose)
5. Serious mental illness or severe Depression assessed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Disorders (SCID-I, DSM-5) and the Montgomery and Asberg Depression Rating Scale (MADRS) scores 24 points or more
6. Clinically significant risk of suicide (Columbia-Suicide Severity Rating Scale (C-SSRC))
7. Women who are pregnant or breastfeeding at screening or Baseline
8. Serious kidney (P-Creatinine > 110 umol/ml) insufficiency
9. The Subject/patient, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason.
10. Liver cirrhosis or liver enzyme elevations, ASAT or ALAT >200 (by blood drop test),
11. Active HCV infection (saliva test, OralQuick-HCV)
12. The person that met the criteria of vulnerable person according to Finnish Medical Research Act No188/1999 7-10§
13. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless surgically sterile must use effective contraception (either combined estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD], intrauterine hormone-releasing system [IUS], vasectomised partner, sexual abstinence (only considered an acceptable method of contraception when it is in line with the subjects' usual and preferred lifestyle), combination of male condom with either cap, diaphragm or sponge with spermicide [double barrier methods]), and willing and able to continue contraception for 1 month after the last administration of IMP. Women using oral contraception must have started using it at least 2 months prior to screening. Women are not considered to be of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms). Or have had a surgical bilateral oophorectomy (with or without hysterectomy) or bilateral tubal ligation at least six weeks before the screening visit. In case of oophorectomy alone, the reproductive status of the woman should have been confirmed by follow up hormone level assessment.
14. Severe comorbidity (e.g., drug addiction, psychosis, diabetes)
15. Experimental agents must have been discontinued at least 8 weeks prior to screening for a period equivalent to 5 half-lives of the agent (whichever is longer)
16. Any diagnosed nasal conditions including abnormal nasal anatomy, nasal symptoms (i.e. blocked nose, nasal polyps etc.), or having product sprayed in to the nasal cavity prior to drug administration
17. Subject with concurrent disease considered by the investigator to be clinically significant in the context of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
The Gambling Symptom Assessment Scale (G-SAS) gambling symptom severity and change during the treatment - assessment | Baseline to week, 3, 6, 9 and week 12.
  The G-SAS is a 12-item self-rated scale designed to assess gambling symptom severity and change during treatment. The G-SAS is not a diagnostic or screening instrument. Each 12-item scale has a score ranging from 0 - 4 (adjective anchors for 0 and 4 vary for each item). All items ask for an average symptom based on the past 7 days. Items 1 - 4 can be used to assess changes in craving symptoms. Total score ranges from 0 - 48: extreme = 41 - 48, severe = 31 - 40, moderate = 21 - 30, mild = 8 - 20.

SECONDARY OUTCOMES:
VAS (gambling craving) | Baseline to Week 3, 6, 9 and 12
  The entire study for an individual participant will last 12 weeks. From baseline to weeks 3,6,9,and 12 craving of gambling will be assessed.
Gambling severity (PGSI) | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. From baseline to weeks 6, and 12 severity of gambling will be assessed.
Gambling severity (DSM-5) | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. From baseline to week 6, and 12 severity of gambling will be assessed.
Gambling problems (NODS) | Baseline to Week 3, 6, 9 and 12
  The entire study for an individual participant will last 12 weeks. From baseline to weeks 3,6,9,and 12 level of gambling problems will be assessed.
Gambling expenditure and frequency | Baseline to Week 12
  daily questionnaire / telephone operated (text messages) diary (daily use of sprays, number of doses, gambling expenditure and frequency and possible adverse events) and self-administration of IMP.
Abstinence of gambling (GASS) | Baseline to Week 3, 6, 9 and 12
  The entire study for an individual participant will last 12 weeks. From baseline to weeks 3,6,9,and 12 abstinence of gambling will be assessed.
Internet use (Internet disorder scale-9 short form) | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. From baseline to weeks 6, and 12 internet use will be assessed.
Quality of life (WHO: EUROHIS-8) | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. From baseline to weeks 6, and 12 quality of life will be assessed.
Alcohol consumption (AUDIT) | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. From baseline to weeks 6, and 12 graving of gambling will be assessed.
Depression (MADRS) | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. From baseline to weeks 6, and 12 mood will be assessed.

OTHER OUTCOMES:
Number and proportion of subjects with adverse events | Baseline to week 12 - daily
  The use of the daily questionnaire / telephone operated (text messages) diary (daily use of sprays, number of doses, gambling expenditure and frequency and possible adverse events) and self-administration of IMP.
Assessment of clinical laboratory parameters - Pregnancy test | Screening to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. At Screening and week 12 blood pregnancy test and week 6 urine pregnancy test
Assessment of vital signs - blood pressure, pulse, temperature | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. Assessments at baseline, 6 and 12 vital signs ( blood pressure, pulse and temperature) will be assessed.
Assessment of body height | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. Assessments at the baseline, week 6, and week 12. Body height will be assessed.
Assessment of body weight | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. Assessment at baseline, 6, and 12 . Body weight will be assessed.
Assessment and examination of nasal mucosa | Baseline to Week 6 and 12
  The entire study for an individual participant will last 12 weeks. Assessment at baseline, 6, and 12 nasal mucosa will be assessed using Nasal Irritation Scale (0= normal appearing mucosa, no bleeding to 5= Ulcerated lesions, bleeding with requires medical intervention). Assessment is performed by MD.
Assessment of smell test | Baseline to Week 12
  The entire study for an individual participant will last 12 weeks. Assessments at baseline and week 12 smell will be assessed.Smell test will be conducted at Baseline and Week 12. NIH Toolbox Odour Identification Test: This validated smell identification test uses 'scratch and sniff' technology, and pictures for the multiple-choice options of 9 common smells. It is intended for a rapid research assessment of olfactory ability.

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Alho, Prof., Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- National Institute for Health and Welfare, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No